CLINICAL TRIAL: NCT01440244
Title: Cervical Video Assisted Thoracoscopic Surgery (C-VATS)Using a Flexible Endoscope for Thoracoscopy
Brief Title: Cervical Video Assisted Thoracoscopic Surgery (C-VATS)
Acronym: CT0030
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 11.092
Record Dates: First submitted 2011-09-16; First posted 2011-09-26 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
Keywords: mediastinoscopy; pleural evaluation; pleural biopsy; pleurodesis
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group assignment (Other): Cervical mediastinoscopy
  Interventions: Procedure: Cervical mediastinoscopy

INTERVENTIONS:
Procedure: Cervical mediastinoscopy — minimally invasive technique to perform pleural evaluation, pleural biopsy and pleurodesis

SUMMARY:
Although thoracic NOTES may not be ready for human trials, a new minimally invasive technique to access the pleural cavity and perform pleural, pulmonary and mediastinal procedures would be possible. Cervical Video Assisted Thoracoscopic Surgery (C-VATS) is a technique that borrows from traditional VATS procedures, from cervical mediastinoscopy, and from flexible endoscopy. All of these procedures are very familiar to the thoracic surgeon.

The current feasibility and safety study examines C-VATS as a method of evaluating, biopsying and performing pleurodesis in patients with pleural disease and or effusion.

DETAILED DESCRIPTION:
Hypothesis: C-VATS is a feasible and safe method of entering the pleural space in order to perform pleural evaluation, pleural biopsy and pleurodesis in patients with pleural disease and/or pleural effusions.

Objectives: Evaluate the safety and feasibility of C-VATS in patients with pleural disease.

Design: Prospective, cohort, feasibility and safety study.

Methods: Patients referred to all thoracic surgeons in the Division of Thoracic Surgery at the CHUM Notre Dame campus for the diagnosis or treatment of pleural based diseases will be screened for enrolment. The investigators plan to recruit 10 patients in this initial study. Eligible patients will be consented by one of the thoracic surgeons at the CHUM.

All procedures will be performing in the operating room at the CHUM Notre Dame Hospital. All patients will be admitted prior to their procedure and treated on the post-operative thoracic surgery ward using standard post-VATS procedural treatments. All cause, as well as procedure specific morbidity will be recorded by the study investigators on the day of the procedure, every day in hospital until discharge and at 1 week, 4 weeks and 12 weeks post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be those that would be candidates for the same pleural procedure (biopsy, drainage and pleurodesis) using a VATS technique

Exclusion Criteria:

* Anticoagulation including Warfarin, Heparin or Clopidogrel which cannot be stopped
* Patients less than 18 years old
* Pregnant patients
* Patient unable to extend neck fully
* Patients with cervical spine instability
* Patients having had previous neck or mediastinal surgery which would preclude mediastinoscopy
* Patients having previously undergone mediastinal irradiation
* Patients having been previously diagnosed with mediastinitis
* Active cervical cutaneous or deep cervical infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
procedure-related morbidity | 30 days
  Intra-operative mortality In-hospital mortality 30-day mortality

SECONDARY OUTCOMES:
pain related to technique | 3-6months
Procedural, hospitalization and overall cost | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada